CLINICAL TRIAL: NCT02346461
Title: An Open-Label Phase 2 Study of ManNAc in Subjects With GNE Myopathy
Brief Title: An Open Label Phase 2 Study of ManNAc in Subjects With GNE Myopathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 150068; 15-HG-0068
Record Dates: First submitted 2015-01-24; First posted 2015-01-27 (Estimated); Results first posted 2019-04-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-03

CONDITIONS: GNE Myopathy
Keywords: Hereditary Inclusion Body Myopathy (HIBM); Sialic Acid (N-acetylneuraminic acid, Neu5Ac); GNE Myopathy; N-Acetyl-D-mannosamine (ManNAc); GNE Gene
MeSH Terms: conditions — Distal myopathy, Nonaka type | interventions — N-acetylmannosamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (2):
- Cohort A (Active Comparator): 6 subjects on Cohort A will receive oral ManNAc 3 g twice daily (6 g/day) for 7 days and, if safe, continue on 6 g twice daily (12 g/day) for the remainder of the study.
  Interventions: Drug: ManNAc
- Cohort B (Active Comparator): 6 subjects on Cohort B will receive oral ManNAc 6 g twice daily (12 g/day) for the duration of the study.
  Interventions: Drug: ManNAc

INTERVENTIONS:
Drug: ManNAc — At doses of 3 g and 6 g twice daily for a total dose of 6 and 12 g per day.
  Arms: Cohort A
Drug: ManNAc — At doses of 6 g twice daily (12 g per day).
  Arms: Cohort B

SUMMARY:
Background:

Patients with GNE myopathy have progressive muscle weakness and can have difficulty walking and decreased mobility. The disease is a rare genetic disorder that results from a gene mutation in a key step in the body's production of a sugar called sialic acid, (also called N-acetylneuraminic acid, Neu5Ac). Researchers think decreased sialic acid bound to muscle proteins may be the cause of muscle wasting in GNE myopathy. Researchers are testing the drug ManNAc which is a precursor in the production of sialic acid within cells. ManNAc is provided as a powder dissolved in water to be administered orally.

DETAILED DESCRIPTION:
GNE myopathy is a rare genetic (autosomal recessive) disorder that causes progressive skeletal muscle atrophy and weakness. The disease presents in young adults typically between the ages of 20 and 40 years, and includes foot drop and difficulty walking. The disease progresses to involve all skeletal muscles, eventually leading to the use of a wheelchair and, in some cases, dependence on a caregiver. The causative gene, GNE, encodes the rate-limiting enzyme in the biosynthesis of CMP-sialic acid. While the exact pathophysiology of GNE myopathy remains unknown, decreased sialic acid production and subsequent hyposialylation of muscle glycoproteins are thought to be key factors leading to muscle deterioration in GNE myopathy. This hypothesis is supported by prevention of disease after administration of oral N-acetyl-D-mannosamine (ManNAc) in mouse models of GNE myopathy. A first-in-human, Phase 1 single ascending dose study evaluated the safety, pharmacokinetics, and pharmacodynamics of a single dose of 3, 6, or 10 g of oral ManNAc in subjects with GNE myopathy (ClinicalTrials.gov NCT01634750; IND No.78,091). ManNAc was safe and well-tolerated in all subjects who participated in this study.

In this Phase 2, open-label, single-center study ManNAc will be administered orally to 12 subjects. The objectives of the study are to assess the long-term safety, tolerability, pharmacokinetics, and biochemical efficacy of oral ManNAc in GNE myopathy subjects. In the first phase of pharmacokinetic assessment, two cohorts of 6 subjects will receive ManNAc at doses of 3 g twice a day (6 g per day) or 6 g twice a day (12 g per day) for 7 days to assess safety and PK. In the second phase of the study, all subjects will receive treatment with ManNAc at a dose of 6 g twice daily (12 g per day) for the remainder of the study. The study was extended to include follow-up evaluations at 6, 12, 18, 24 and 30 months. During the 30 month visit, PK of 4 g three times daily was assessed. Biochemical efficacy was assessed by change in the sialylation of proteins at 3 months compared to baseline. To evaluate the effect of ManNAc on clinical measures of GNE myopathy, a battery of clinical assessments was performed at every visit to identify clinical endpoints suitable for subsequent clinical trials.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Subject is age 18-60 years, inclusive, and of either gender.
* Subject has a diagnosis of GNE myopathy based upon a consistent clinical course and identification of two GNE gene mutations.
* Subject must be willing to stop any treatment with ManNAc, sialic acid, intravenous immunoglobulin (IVIG), and/or other supplements containing sialic acid (e.g. St. John s wort, sialyllactose) 90 days prior to dosing and remain off such treatment for the duration of the trial.
* Subjects must have a body mass index (BMI) between 18 and 30 kg/m2, with a bodyweight of >50 kg.
* Subjects must have 20-75% of predicted strength measured by QMA at baseline on at least one of the following: 1) ankle dorsiflexion, 2) knee flexion, 3) hip extension, 4) grip, 5) elbow flexion, shoulder abduction

  * 20-75% of predicted strength measures by OMA at baseline, or
  * If predicted muscle strength above 75%, a documented change of at least 10% per year.
* Subject has the ability to travel to the NIH Clinical Center for admissions.
* Subject has an INR less than or equal to 1.5 and must have stopped warfarin and other anticoagulants 2 weeks prior and after muscle biopsy procedures. Aspirin and clopidogrel should be stopped 3 days and 5 days before the procedure, respectively.
* Subject must be able to comply with requirements of the protocol, including blood collection, drug administration, muscle MRI/MRS, muscle biopsy and muscle strength assessments.
* If a woman of reproductive age, subject must be willing to use an effective method of contraception for the duration of the trial.
* Subject must be able to provide informed consent.

EXCLUSION CRITERIA:

* Subject had a clinical significant infection or medical illness 30 days prior to the first protocol visit.
* Subject has a psychiatric illness or neurological disease that would interfere with the ability to comply with the requirements of this protocol. This includes, but is not limited to, uncontrolled/untreated psychotic depression, bipolar disorder, schizophrenia, substance abuse or dependence, antisocial personality disorder, panic disorder, or behavioral problems, which interfere with effective communication.
* Subject has hepatic laboratory parameters (AST, ALT, GGTP) or renal laboratory parameters (creatinine, BUN) greater than 3 times the upper limit of normal.
* Subject has known adverse reactions to anesthetic or sedatives utilized for muscle biopsy.
* Subject is anemic (defined as Hematocrit <30%) or has platelets <100,000 or white blood cell count less than 3,000.
* Subject shows evidence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematological, metabolic, or gastrointestinal disease, or has a condition that requires immediate surgical intervention.
* Subject is pregnant or breastfeeding at any time during the study.
* Subject has received treatment with another investigational drug, investigational device, or approved therapy for investigational use less than 90 days prior to the first protocol visit.
* Subject has hypersensitivity to ManNAc or in the judgment of the investigator, has a condition that places the subject at increased risk for adverse effects.
* Subject has received ManNAc, sialic acid, intravenous immunoglobulin (IVIG), and/or other supplements containing sialic acid (e.g. St. John s wort, sialyllactose) less than 90 days prior to the first protocol visit.
* The presence of persistent diarrhea or malabsorption that could interfere with the subject s ability to absorb drugs or to tolerate ManNAc therapy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2015-02-05 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2018-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nuria Carrillo, M.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Carrillo N, Malicdan MC, Leoyklang P, Shrader JA, Joe G, Slota C, Perreault J, Heiss JD, Class B, Liu CY, Bradley K, Jodarski C, Ciccone C, Driscoll C, Parks R, Van Wart S, Bayman L, Coffey CS, Quintana M, Berry SM, Huizing M, Gahl WA. Safety and efficacy of N-acetylmannosamine (ManNAc) in patients with GNE myopathy: an open-label phase 2 study. Genet Med. 2021 Nov;23(11):2067-2075. doi: 10.1038/s41436-021-01259-x. Epub 2021 Jul 13. PMID 34257421
- [Derived] Van Wart S, Mager DE, Bednasz CJ, Huizing M, Carrillo N. Population Pharmacokinetic Model of N-acetylmannosamine (ManNAc) and N-acetylneuraminic acid (Neu5Ac) in Subjects with GNE Myopathy. Drugs R D. 2021 Jun;21(2):189-202. doi: 10.1007/s40268-021-00343-6. Epub 2021 Apr 24. PMID 33893973

RESULTS

PARTICIPANT FLOW:
Groups:
- ManNAc: Cohort A: Cohort A received oral ManNAc 3 g twice daily (6 g/day) for 7 days and, then were escalated to 6 g twice daily (12 g/day) for the remainder of the study.
- ManNAc: Cohort B: Cohort B received oral ManNAc 6 g twice daily (12 g/day) for the duration of the study.
Period: Overall Study
Arm/Group | ManNAc: Cohort A | ManNAc: Cohort B
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ManNAc: Cohort A | ManNAc: Cohort B | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 12
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 2 | 4 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 6 | 12
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 4 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Area Under the Curve (AUClast) of Plasma ManNAc (Baseline-adjusted)
Description: The mean area under the plasma ManNAc concentration-versus time curve from time 0 (dosing) to the time of last quantifiable concentration.
Time Frame: Day 7
Population: All subjects received ManNAc
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Groups:
- ManNAc: Cohort A: ManNAc 3 g twice daily (6 g/day) for 7 days
- ManNAc: Cohort B: ManNAc 6 g twice daily (12 g/day)
Arm/Group | ManNAc: Cohort A | ManNAc: Cohort B
Number analyzed (Participants) | 6 | 6
hr*ng/mL | 7461 (1776) | 9432 (2710)

2. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of ManNAc (Baseline-adjusted)
Description: The maximum (or peak) plasma ManNAc concentration that the drug achieves in the body after the drug has been administrated.
Time Frame: Day 7
Population: All subjects received ManNAc
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | ManNAc: Cohort A | ManNAc: Cohort B
Number analyzed (Participants) | 6 | 6
ng/mL | 1588 (28.9) | 1774 (21.2)

3. Primary Outcome: The Time to Cmax (Tmax) for ManNAc
Description: The time taken to achieve the maximum observed plasma concentration for ManNAc .
Time Frame: Day 7
Population: All subjects received ManNAc
Measure: Median (Standard Deviation); unit: hours
Arm/Group | ManNAc: Cohort A | ManNAc: Cohort B
Number analyzed (Participants) | 6 | 6
hours | 2.0 (0.4) | 2.5 (0.8)

4. Primary Outcome: Half-life (t ½) for ManNAc
Description: The amount of time it takes for plasma ManNAc concentration to decline by half.
Time Frame: Day 7
Population: All subjects received ManNAc
Measure: Median (Standard Deviation); unit: hours
Arm/Group | ManNAc: Cohort A | ManNAc: Cohort B
Number analyzed (Participants) | 6 | 6
hours | 2.0 (0.3) | 2.1 (1.1)

5. Primary Outcome: Mean Area Under the Curve (AUClast) of Plasma Neu5Ac (Baseline-adjusted)
Description: The mean area under the plasma Neu5Ac concentration-versus time curve from time 0 (dosing) to the time of last quantifiable concentration.
Time Frame: Day 7
Population: All subjects received ManNAc
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | ManNAc: Cohort A | ManNAc: Cohort B
Number analyzed (Participants) | 6 | 6
hr*ng/mL | 4206 (1352) | 5175 (1421)

6. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Neu5Ac (Baseline-adjusted)
Description: The maximum (or peak) plasma Neu5Ac concentration that the drug achieves in the body after the drug has been administrated.
Time Frame: Day 7
Population: All subjects received ManNAc
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | ManNAc: Cohort A | ManNAc: Cohort B
Number analyzed (Participants) | 6 | 6
ng/mL | 469 (35.1) | 620 (25.5)

7. Primary Outcome: The Time to Cmax (Tmax) for Neu5Ac
Description: The time taken to achieve the maximum observed plasma concentration for Neu5Ac.
Time Frame: Day 7
Population: All subjects received ManNAc
Measure: Median (Standard Deviation); unit: hours
Arm/Group | ManNAc: Cohort A | ManNAc: Cohort B
Number analyzed (Participants) | 6 | 6
hours | 8.0 (4.1) | 6.0 (3.4)

ADVERSE EVENTS:
Time Frame: 30 months
Groups:
- ManNAc 3 g - 7 Days: Subjects who received oral ManNAc 3 g twice daily (6 g/day) for the first 7 days.
- ManNAc 6 g - 7 Days: Subjects who received oral ManNAc 6 g twice daily (12 g/day) for the first 7 days.
- ManNAc 6 g - Day 8 to 30 Months: All subjects received oral ManNAc 6 g twice daily (12 g/day) from day 8 to the end of the study at 30 months.
Arm/Group | ManNAc 3 g - 7 Days | ManNAc 6 g - 7 Days | ManNAc 6 g - Day 8 to 30 Months
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/12
Other Adverse Events (participants affected / at risk) | 5/6 | 6/6 | 12/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ManNAc 3 g - 7 Days (N=6) | ManNAc 6 g - 7 Days (N=6) | ManNAc 6 g - Day 8 to 30 Months (N=12)
Abdominal distension (Gastrointestinal disorders) | 2 | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 2 | 7
Alanine aminotransferase increased (Investigations) | 2 | 3 | 6
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 3
Aspartate aminotransferase increased (Investigations) | 1 | 4 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Basal cell carcinoma (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1 | 1
Blood cholesterol increased (Investigations) | 0 | 0 | 3
Blood creatine phosphokinase increased (Investigations) | 2 | 4 | 8
Bronchitis (Infections and infestations) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 3
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 2
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 5
Flatulence (Gastrointestinal disorders) | 2 | 2 | 4
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 2
Haematuria (Renal and urinary disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 5
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 | 0 | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Obesity (Metabolism and nutrition disorders) | 2 | 0 | 6
Oedema peripheral (General disorders) | 1 | 0 | 0
Pain (General disorders) | 1 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 2
Sinusitis (Infections and infestations) | 0 | 0 | 1
Skin induration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 2
syncope (Nervous system disorders) | 0 | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 2
Weight decreased (Investigations) | 0 | 0 | 1
Weight increased (Investigations) | 0 | 0 | 5
White blood cell count decreased (Investigations) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-07): https://cdn.clinicaltrials.gov/large-docs/61/NCT02346461/Prot_SAP_000.pdf